CLINICAL TRIAL: NCT01516723
Title: Hybrid Sirolimus-eluting Stent With Bioresorbable Polymer Versus Everolimus-eluting Stent With Durable Polymer for Total Coronary Occlusions in Native Coronary Arteries (PRISON-IV)
Brief Title: Hybrid Sirolimus-eluting Versus Everolimus-eluting Stents for Total Coronary Occlusions
Acronym: PRISON-IV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: R&D Cardiologie (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Dr. M.J. Suttorp, MD, PhD, R&D Cardiologie
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDC-2011-02
Record Dates: First submitted 2011-11-15; First posted 2012-01-25 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease; Coronary Disease; Coronary Stenosis
Keywords: drug-eluting stent; chronic total occlusion; hybrid sirolimus-eluting stent; everolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid sirolimus-eluting stents (Experimental): ORSIRO, Biotronik Inc.
  Interventions: Device: Hybrid sirolimus- and everolimus-eluting stents (ORSIRO, XIENCE PRIME)
- Everolimus-eluting stents (Active Comparator): XIENCE PRIME, Abbott
  Interventions: Device: Hybrid sirolimus- and everolimus-eluting stents (ORSIRO, XIENCE PRIME)

INTERVENTIONS:
Device: Hybrid sirolimus- and everolimus-eluting stents (ORSIRO, XIENCE PRIME) — Recanalization of totally occluded coronary arteries
  Other Names: Hybrid sirolimus-eluting stents (ORSIRO, Biotronik); Everolimus-eluting stents (XIENCE PRIME, Abbott)

SUMMARY:
Percutaneous recanalization of total coronary occlusions (TCO) was historically hampered by high rates of restenosis and reocclusion. In the PRISON II and III trial we showed landmark reduction in restenosis with sirolimus-eluting stents (Cypher, Cordis Corporation) compared to conventional bare metal stents in TCO. In the PRISON III trial, we observed similar favourable results with second-generation zotarolimus-eluting stent (Resolute, Medtronic Inc.). Another drugs-eluting stent mounted with everolimus (Xience Prime, Abbott) also demonstrated favourable results in TCO. Recently, drug-eluting stents (DES) with bioresorbable polymer coatings were developed, to address safety concerns regarding the observation of very late stent thrombosis, due to hypersensitivity reactions, and chronic inflammation, on the durable polymer coating of DES. However, none of these DES with bioresorbable polymers were evaluated in patients with TCO. The PRISON IV trial is a prospective, randomized, single-blinded, multi-center trial, designed to evaluate the safety, efficacy, and angiographic outcome of hybrid sirolimus-eluting stents with bioresorbable polymers (ORSIRO, Biotronik Inc.) compared to everolimus-eluting stents with durable polymers (Xience Prime, Abbott) in patients with successfully recanalized TCOs.

DETAILED DESCRIPTION:
A total of 330 patients are randomized to either hybrid sirolimus-eluting stent or everolimus-eluting stent after successful recanalization of TCO. Clinical follow-up at 1, 6, 12 months, 2, 3, 4, 5 year with angiographic follow-up at 9 months. In 60 patients a optical coherence tomography is performed during the 9 months follow-up angiography. Quantitative coronary and optical coherence tomography analysis is performed by two independent core laboratory. The primary end point is in-segment late luminal loss at 9 month angiographic follow-up. Secondary angiographic end points include the following; in-stent luminal loss, acute recoil, acute gain, net luminal gain, late loss index, minimal lumen diameter, percentage of diameter stenosis, in-stent and in-segment binary restenosis and reocclusions at 9 months angiographic follow-up. Secondary clinical endpoints include a composite of major adverse cardiac events (death, MI and clinically driven target lesion revascularization); clinically driven target vessel revascularisation (TVR), target vessel failure (cardiac death, MI, clinically driven TVR) and stent thrombosis up to 5 year clinical follow-up. Tertiary optical coherence tomography end points at 9 months follow-up are the following: Percentage of uncovered stent struts, percentage of malapposed stent struts, tissue strut thickness, absolute and percentage of intimal hyperplasia.

ELIGIBILITY:
INCLUSION CRITERIA:

* the estimated duration of the occlusion is at least 4 weeks.
* signs of ischemia related to the occluded coronary artery.
* successful recanalization of the occluded artery is achieved.
* reference diameter is > 2.5 mm.
* written informed consent obtained.

EXCLUSION CRITERIA:

* primary or rescue PCI for acute myocardial infarction
* the lesion could not be crossed.
* lesions with complex anatomy making successful stent deployment unlikely.
* the guide wire is not in the true lumen distal to the occlusion.
* Sirolimus or zotarolimus allergy
* venous or arterial bypass grafts
* pregnant or nursing women.
* participation in an other trial.
* factors making long-term follow-up difficult or unlikely.
* life expectancy < 1 year.
* contraindications for ASA or Clopidogrel or heparin.
* use of coumadins that could not be stopped before the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
In-segment late luminal loss at 9 months as assessed by an independent angiographic core lab. | 9 month

SECONDARY OUTCOMES:
In-stent late luminal loss | 9 month
In-stent and in-segment binary restenosis rate | 9 month
In-stent and in-segment minimal lumen diameter | 9 month
Percentage diameter stenosis | 9 month
A composite of major adverse cardiac events (MACE: death, myocardial infarction and clinically driven target lesion revascularization) | 9 month
Stent thrombosis (acute, <1day; subacute, 1 to 30 days; and late, >30 days) | 30 days
Target vessel failure (cardiac death, MI, clinically driven target vessel revascularisation) up to 5 year of clinical follow-up. | 5 years
% of uncovered stent struts, % of malapposed stent struts, tissue strut thickness (µm), absolute volume (mm³) and % of intimal hyperplasia | 9 month
  Assessed by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Maarten J. Suttorp, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (4):
- AZ Middelheim, Antwerp, Antwerpen, Belgium
- Netherlands (3):
  - AMC, Amsterdam, Amsterdam
  - Catharina Ziekenhuis, Eindhoven, Eindhoven
  - St Antonius Hospital, Nieuwegein

REFERENCES:
- [Background] Rahel BM, Suttorp MJ, Laarman GJ, Kiemeneij F, Bal ET, Rensing BJ, Ernst SM, ten Berg JM, Kelder JC, Plokker HW. Primary stenting of occluded native coronary arteries: final results of the Primary Stenting of Occluded Native Coronary Arteries (PRISON) study. Am Heart J. 2004 May;147(5):e22. doi: 10.1016/j.ahj.2003.11.023. PMID 15131557
- [Background] Suttorp MJ, Mast EG, Plokker HW, Kelder JC, Ernst SM, Bal ET. Primary coronary stenting after successful balloon angioplasty of chronic total occlusions: a single-center experience. Am Heart J. 1998 Feb;135(2 Pt 1):318-22. doi: 10.1016/s0002-8703(98)70099-7. PMID 9489982
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Sirnes PA, Golf S, Myreng Y, Molstad P, Emanuelsson H, Albertsson P, Brekke M, Mangschau A, Endresen K, Kjekshus J. Stenting in Chronic Coronary Occlusion (SICCO): a randomized, controlled trial of adding stent implantation after successful angioplasty. J Am Coll Cardiol. 1996 Nov 15;28(6):1444-51. doi: 10.1016/s0735-1097(96)00349-x. PMID 8917256
- [Background] Suttorp MJ, Laarman GJ, Rahel BM, Kelder JC, Bosschaert MA, Kiemeneij F, Ten Berg JM, Bal ET, Rensing BJ, Eefting FD, Mast EG. Primary Stenting of Totally Occluded Native Coronary Arteries II (PRISON II): a randomized comparison of bare metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions. Circulation. 2006 Aug 29;114(9):921-8. doi: 10.1161/CIRCULATIONAHA.106.613588. Epub 2006 Aug 14. PMID 16908768
- [Background] Kandzari DE, Leon MB, Popma JJ, Fitzgerald PJ, O'Shaughnessy C, Ball MW, Turco M, Applegate RJ, Gurbel PA, Midei MG, Badre SS, Mauri L, Thompson KP, LeNarz LA, Kuntz RE; ENDEAVOR III Investigators. Comparison of zotarolimus-eluting and sirolimus-eluting stents in patients with native coronary artery disease: a randomized controlled trial. J Am Coll Cardiol. 2006 Dec 19;48(12):2440-7. doi: 10.1016/j.jacc.2006.08.035. Epub 2006 Nov 28. PMID 17174180
- [Background] Wohrle J, Rottbauer W, Imhof A. Everolimus-eluting stents for treatment of chronic total coronary occlusions. Clin Res Cardiol. 2012 Jan;101(1):23-8. doi: 10.1007/s00392-011-0359-3. Epub 2011 Sep 22. PMID 21938564
- [Background] Rahel BM, Laarman GJ, Kelder JC, Ten Berg JM, Suttorp MJ. Three-year clinical outcome after primary stenting of totally occluded native coronary arteries: a randomized comparison of bare-metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions (Primary Stenting of Totally Occluded Native Coronary Arteries [PRISON] II study). Am Heart J. 2009 Jan;157(1):149-55. doi: 10.1016/j.ahj.2008.08.025. Epub 2008 Nov 6. PMID 19081412
- [Background] Van den Branden BJ, Rahel BM, Laarman GJ, Slagboom T, Kelder JC, Ten Berg JM, Suttorp MJ. Five-year clinical outcome after primary stenting of totally occluded native coronary arteries: a randomised comparison of bare metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions (PRISON II study). EuroIntervention. 2012 Feb;7(10):1189-96. doi: 10.4244/EIJV7I10A190. PMID 22030323
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Background] Virmani R, Liistro F, Stankovic G, Di Mario C, Montorfano M, Farb A, Kolodgie FD, Colombo A. Mechanism of late in-stent restenosis after implantation of a paclitaxel derivate-eluting polymer stent system in humans. Circulation. 2002 Nov 19;106(21):2649-51. doi: 10.1161/01.cir.0000041632.02514.14. PMID 12438288
- [Background] Cook S, Ladich E, Nakazawa G, Eshtehardi P, Neidhart M, Vogel R, Togni M, Wenaweser P, Billinger M, Seiler C, Gay S, Meier B, Pichler WJ, Juni P, Virmani R, Windecker S. Correlation of intravascular ultrasound findings with histopathological analysis of thrombus aspirates in patients with very late drug-eluting stent thrombosis. Circulation. 2009 Aug 4;120(5):391-9. doi: 10.1161/CIRCULATIONAHA.109.854398. Epub 2009 Jul 20. PMID 19620501
- [Background] Stefanini GG, Kalesan B, Serruys PW, Heg D, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Wijns W, Morice MC, Di Mario C, Corti R, Antoni D, Sohn HY, Eerdmans P, van Es GA, Meier B, Windecker S, Juni P. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer sirolimus-eluting stents in patients with coronary artery disease (LEADERS): 4 year follow-up of a randomised non-inferiority trial. Lancet. 2011 Dec 3;378(9807):1940-8. doi: 10.1016/S0140-6736(11)61672-3. Epub 2011 Nov 8. PMID 22075451
- [Background] Ughi GJ, Adriaenssens T, Onsea K, Kayaert P, Dubois C, Sinnaeve P, Coosemans M, Desmet W, D'hooge J. Automatic segmentation of in-vivo intra-coronary optical coherence tomography images to assess stent strut apposition and coverage. Int J Cardiovasc Imaging. 2012 Feb;28(2):229-41. doi: 10.1007/s10554-011-9824-3. Epub 2011 Feb 24. PMID 21347593
- [Background] Moreno R, Garcia E, Teles RC, Almeida MS, Carvalho HC, Sabate M, Martin-Reyes R, Rumoroso JR, Galeote G, Goicolea FJ, Moreu J, Mainar V, Mauri J, Ferreira R, Valdes M, Perez de Prado A, Martin-Yuste V, Jimenez-Valero S, Sanchez-Recalde A, Calvo L, Lopez de Sa E, Macaya C, Lopez-Sendon JL. A randomised comparison between everolimus-eluting stent and sirolimus-eluting stent in chronic coronary total occlusions. Rationale and design of the CIBELES (non-acute Coronary occlusion treated by EveroLimus-Eluting Stent) trial. EuroIntervention. 2010 May;6(1):112-6. PMID 20542806
- [Derived] Teeuwen K, Adriaenssens T, Van den Branden BJ, Henriques JP, Van der Schaaf RJ, Koolen JJ, Vermeersch PH, Bosschaert MA, Tijssen JG, Suttorp MJ. A randomized multicenter comparison of hybrid sirolimus-eluting stents with bioresorbable polymer versus everolimus-eluting stents with durable polymer in total coronary occlusion: rationale and design of the Primary Stenting of Occluded Native Coronary Arteries IV study. Trials. 2012 Dec 15;13:240. doi: 10.1186/1745-6215-13-240. PMID 23241457